CLINICAL TRIAL: NCT04169581
Title: Symmetricity-Driven Learning Framework for Pediatric Temporal Lobe Epilepsy Detection Using 18F-FDG-PET Imaging
Brief Title: A Deep Learning Framework for Pediatric TLE Detection Using 18F-FDG-PET Imaging
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-124
Record Dates: First submitted 2019-11-13; First posted 2019-11-20 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-06

CONDITIONS: Epilepsy, Temporal Lobe
Keywords: Deep Learning; Temporal Lobe Epilepsy; Positron-Emission Tomography
MeSH Terms: conditions — Epilepsy, Temporal Lobe

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: The experimental group received 18F-FDG PET examination
- Control Group: The control group received 18F-FDG PET examination

SUMMARY:
This study aims to use radiomics analysis and deep learning approaches for seizure focus detection in pediatric patients with temporal lobe epilepsy (TLE). Ten positron emission tomograph (PET) radiomics features related to pediatric temporal bole epilepsy are extracted and modelled, and the Siamese network is trained to automatically locate epileptogenic zones for assistance of diagnosis.

DETAILED DESCRIPTION:
Purpose:The key to successful epilepsy control involves locating epileptogenic focus before treatment. 18F-FDG PET has been considered as a powerful neuroimaging technology used by physicians to assess patients for epilepsy. However, imaging quality, viewing angles, and experiences may easily degrade the consistency in epilepsy diagnosis. In this work, the investigators develop a framework that combines radiomics analysis and deep learning techniques to a computer-assisted diagnosis (CAD) method to detect epileptic foci of pediatric patients with temporal lobe epilepsy (TLE) using PET images.

Methods:Ten PET radiomics features related to pediatric temporal bole epilepsy are first extracted and modelled. Then a neural network called Siamese network is trained to quanti-fy the asymmetricity and automatically locate epileptic focus for diagnosis.The performance of the proposed framework was tested and compared with both the state-of-art clinician software tool and human physicians with different levels of experiences to validate the accuracy and consistency.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of temporal lobe epilepsy.
2. Age range from six to eighteen years old.
3. Underwent PET, EEG, computed tomography (CT) and MRI.

Exclusion Criteria:

1. Image quality is unsatisfactory (e.g. severe image artifacts due to head movement).
2. 18F-FDG PEG examination is negative.
3. Clinical data is incomplete.
4. EEG or MRI report is missing.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with Temporal Lobe Epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
The 'area under curve' (AUC ) of our model in detection performance | Through study completion, about 1 year
  To evaluate the performance of our model, the investigators calculated the AUC of our model for normal or abnormal classification campared with different methods and and physicians with different levels.

SECONDARY OUTCOMES:
The 'dice similarity coefficient' (DSC) of our model in detection performance | Through study completion, about 3 months
  The accuracy of focus lesion detection is quantitatively measured through the metric of 'dice similarity coefficient' (DSC) by comparing the spatial overlap between the marked regions between the reference standard and the subject method under test.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine and PET/CT Center, The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Q, Liao Y, Wang X, Zhang T, Feng J, Deng J, Shi K, Chen L, Feng L, Ma M, Xue L, Hou H, Dou X, Yu C, Ren L, Ding Y, Chen Y, Wu S, Chen Z, Zhang H, Zhuo C, Tian M. A deep learning framework for 18F-FDG PET imaging diagnosis in pediatric patients with temporal lobe epilepsy. Eur J Nucl Med Mol Imaging. 2021 Jul;48(8):2476-2485. doi: 10.1007/s00259-020-05108-y. Epub 2021 Jan 9. PMID 33420912